CLINICAL TRIAL: NCT02250417
Title: Investigation of a Novel Sleep Surface for Treatment of Positional Sleep Apnea.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Hill-Rom (Industry)
Responsible Party: Principal Investigator, Ulysses Magalang MD, Professor of Medicine, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2014H0235
Record Dates: First submitted 2014-09-23; First posted 2014-09-26 (Estimated); Results first posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wave Surface, Then Non Wave Surface (Experimental): Subjects sleep first for a whole night in the sleep laboratory with the Wave sleep surface. They then return to the sleep laboratory and sleep without the Wave sleep surface.
  Interventions: Other: Wave sleep surface
- Non Wave Surface, Then Wave Surface (Experimental): Subjects sleep first for a whole night in the sleep laboratory without the Wave sleep surface. They then return to the sleep laboratory and sleep with the Wave sleep surface.
  Interventions: Other: Wave sleep surface

INTERVENTIONS:
Other: Wave sleep surface — The Wave sleep surface is designed to be used as a bed surface and with any combinations of sleep pillows, bed linens, and bed clothes and intended to avoid the supine position during sleep.

SUMMARY:
Body position during sleep influences the severity of obstructive sleep apnea (OSA). The AHI is the number of times per hour of sleep that the airway temporarily collapses at the level of the tongue or soft palate. In a significant number of individuals with OSA, the severity of the condition as measured by the apnea-hypopnea index (AHI), increases in the supine (back) position and lowers in the lateral (side) position. This is called positional OSA.

The primary objective of this study is to determine whether sleeping with a novel sleep surface (Wave sleep surface) that is used on top of a regular bed reduces the AHI in those with positional OSA.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether sleeping with the novel device (Wave sleep surface) reduces the AHI in those with supine position-related OSA, also known as positional OSA. A secondary aim is to determine the effects of the sleep surface on subjective and objective measures of sleep in patients with positional OSA.

ELIGIBILITY:
Inclusion Criteria:

We will recruit subjects who are:

* 18 years of age and above
* Willing and able to give informed consent
* Prior sleep study done based on previous clinical evaluation by the subject's treating physician in the course of usual clinical care and performed no more than 12 months prior to enrollment that meets the following:

  * overall AHI 5-30 events/hr
  * at least 20 minutes of recorded sleep in the supine and nonsupine postures
  * positional OSA defined as > 50% reduction in the AHI between the supine and nonsupine postures and AHI < 5hr in the nonsupine position
  * central apneas < 50% of the total number of apneas and hypopneas
* Patients who meet the above criteria who have been prescribed CPAP therapy but are non-compliant will be enrolled in the study. CPAP noncompliance will be defined as average nightly use < 4hrs/night based on a download of the CPAP machine, or self- acknowledged discontinuation of CPAP use.

Exclusion Criteria:

* Incapable of giving informed consent
* Under the age of 18
* Known inability to sleep in the lateral position
* Active titration of medication
* Excessive alcohol consumption

  * Excessive alcohol use is defined as:
  * More than 3 glasses of wine a day
  * More than 3 beers a day
  * More than 60 mL of hard liquor a day
* Room air oxyhemoglobin saturation < 88%
* Use of home oxygen
* Compliant with OSA therapy
* Presence of severe daytime sleepiness defined as an Epworth sleepiness scale score > 16 or a prior history of falling asleep while driving
* Unstable medical problem such as uncontrolled hypertension.
* Body Mass Index (BMI) > 45 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-08; Primary Completion 2015-04 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulysses J Magalang, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Martha Morehouse Medical Pavilion 2050 Kenny Rd;Ste 2600, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Participants randomized to Wave Sleep Surface, then to Non Wave Surface
- Sequence 2: Participants randomized to Non Wave Sleep Surface, then to the Wave Sleep Surface
Period: First Intervention (1 Night)
Arm/Group | Sequence 1 | Sequence 2
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Second Intervention (1 Night)
Arm/Group | Sequence 1 | Sequence 2
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This is a randomized cross-over study. The same subject slept with and without the Wave sleep surface.
Groups:
- All Study Participanrts: Participants with positional OSA (based on a previously performed baseline clinical study) were randomized to sleep with or without the Wave sleep surface in a cross-over design. Baseline PSG measures represent values from the previously performed clinical study that qualified subjects to have positional OSA.
Arm/Group | All Study Participanrts
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 12
Total AHI [Mean (Standard Deviation); unit: events/hr] | 14.4 (5.8)
supine AHI [Mean (Standard Deviation); unit: events/hr] | 38.1 (24.6)
non-supine AHI [Mean (Standard Deviation); unit: events/hr] | 1.6 (1.1)
Total Sleep Time [Mean (Standard Deviation); unit: mins] | 364.5 (43.8)
Total Recording Time [Mean (Standard Deviation); unit: mins] | 415.7 (32.0)
Sleep Efficiency [Mean (Standard Deviation); unit: %] — Sleep Efficiency=total sleep time divided by total recording time x100
  % | 87.6 (7.2)
Supine Sleep Time [Mean (Standard Deviation); unit: mins] | 153.8 (84.7)
Non-supine Sleep Time [Mean (Standard Deviation); unit: mins] | 210.7 (79.7)
Stage N1 Duration [Mean (Standard Deviation); unit: minutes] — Stage N1 is the lightest sleep stage
  minutes | 33.3 (17.0)
Stage N2 Duration [Mean (Standard Deviation); unit: minutes] — Stage N2 Duration is referred to as the longest sleep stage/largest percentage of sleep time
  minutes | 255.8 (48.8)
Stage N3 Duration [Mean (Standard Deviation); unit: minutes] — Stage N3 is the referred to as "deep sleep" or "slow wave sleep."
  minutes | 21.1 (23.0)
Stage R Duration [Mean (Standard Deviation); unit: minutes] — Stage R is the last sleep stage-rapid eye movement (REM)
  minutes | 50.8 (30.1)

OUTCOME MEASURES:

1. Primary Outcome: Apnea-hypopnea Index (AHI)- Intention to Treat Analysis
Description: AHI, or the apnea-hypopnea index, is a numerical measure that accounts for the number of pauses in your breathing per hour of sleep.
  These breathing disturbances are typically associated with either a brief arousal or awakening from sleep or a 4 percent drop in the blood oxygen levels, called a desaturation. It is used to assess the severity of an individual's sleep apnea.
  This is measured in each study participant when sleeping with the Wave Sleep Surface and sleeping without the Wave Sleep Surface.
Time Frame: measured during each of the two sleep study sessions (Study Visits 2 and 3)
Population: The study compares the difference in AHI within each study subject with and without the use of the Wave Sleep Surface during visit 2 and 3 (intention to treat analysis).
Measure: Mean (Standard Deviation); unit: events/hr
Groups:
- Wave Night: Results of PSG while sleeping in the sleep laboratory with the Wave sleep surface.
- Non-Wave Night: Results of PSG while sleeping in the sleep laboratory without the Wave sleep surface.
Arm/Group | Wave Night | Non-Wave Night
Number analyzed (Participants) | 12 | 12
events/hr | 9.8 (9.4) | 12.6 (7.3)

2. Secondary Outcome: Objective Sleep Quality
Description: Sleep quality assessment using objective sleep architecture measures during PSG performed during the non-Wave Sleep Surface night compared to the Wave Sleep Surface night during visits 2 and 3.
Time Frame: measured during each of the two sleep study sessions (Study Visits 2 and 3)
Population: Intention to treat analysis includes data from non-wave night regardless of time spent in supine position compared to baseline polysomnography.
Measure: Mean (Standard Deviation); unit: mins
Arm/Group | Non-Wave Night | Wave Night
Number analyzed (Participants) | 12 | 12
mins
  Total Sleep Time | 379.8 (31.9) | 363.7 (23.8)
  Total Recording Time | 424.1 (34.5) | 414.3 (24.2)
  Stage N1 duration(lightest sleep stage) | 38.8 (19.1) | 36.5 (17.9)
  Stage N2 duration(longest sleep stage) | 261.8 (34.8) | 259.3 (19.5)
  StageN3 duration(deep sleep stage) | 14.1 (16.0) | 14.8 (16.2)
  Stage R duration(Rapid eye movement or REM) | 65.0 (23.1) | 53.1 (34.7)

3. Post Hoc Outcome: Apnea-hypopnea Index (AHI)- Modified Analysis
Description: AHI, or the apnea-hypopnea index, is a numerical measure that accounts for the number of pauses in breathing per hour of sleep.
  These breathing disturbances are typically associated with either a brief arousal or awakening from sleep or a 4 percent drop in the blood oxygen levels, called a desaturation. It is used to assess the severity of an individual's sleep apnea.
  This is measured in each study participant when sleeping with the Wave Sleep Surface and sleeping without the Wave Sleep Surface.
  The modified analysis compares the AHI within each participant where time spent in the supine position is greater than time spent in non-supine position from either the baseline (inclusion) sleep study or the non-Wave night sleep study compared to the Wave Sleep Surface night sleep study.
Time Frame: Baseline (inclusion) sleep study or the non-Wave night sleep study compared to the Wave Sleep Surface night sleep study.
Population: Modified analysis compares the AHI when the time spent in supine position is greater than in the non-supine position either during the baseline sleep study or the non-Wave night.The baseline PSG is the clinical PSG that was the basis of the inclusion to the study performed prior to randomization.
Measure: Mean (Standard Deviation); unit: events/hr
Groups:
- Non-Wave Night: Results of PSG while sleeping in the sleep laboratory without the Wave sleep surface when the time spent in supine position is greater than time spent in non-supine position either during the baseline (inclusion) PSG study or the Non-Wave Sleep Surface night PSG.
  The baseline PSG is the clinical PSG that was the basis of the inclusion to the study performed prior to randomization.
Arm/Group | Wave Night | Non-Wave Night
Number analyzed (Participants) | 12 | 12
events/hr | 9.8 (9.4) | 15.9 (6.4)

4. Secondary Outcome: Sleep Efficiency
Description: Sleep quality assessment using objective sleep architecture measures during PSG performed during the non-Wave Sleep Surface night compared to the Wave Sleep Surface night during visits 2 and 3. Sleep efficiency is defined as the total sleep time divided by the total recording time X100.
Time Frame: measured during each of the two sleep study sessions (Study Visits 2 and 3)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of total recording time
Arm/Group | Non-Wave Night | Wave Night
Number analyzed (Participants) | 12 | 12
percentage of total recording time | 89.9 (7.8) | 87.9 (5.6)

ADVERSE EVENTS:
Time Frame: 7 months
Groups:
- Sequence 1: Subjects sleep first for a whole night in the sleep laboratory with the Wave sleep surface. They then return to the sleep laboratory and sleep without the Wave sleep surface.
  Wave sleep surface: The Wave sleep surface is designed to be used as a bed surface and with any combinations of sleep pillows, bed linens, and bed clothes and intended to avoid the supine position during sleep.
- Sequence 2: Subjects sleep first for a whole night in the sleep laboratory without the Wave sleep surface. They then return to the sleep laboratory and sleep with the Wave sleep surface.
  Wave sleep surface: The Wave sleep surface is designed to be used as a bed surface and with any combinations of sleep pillows, bed linens, and bed clothes and intended to avoid the supine position during sleep.
Arm/Group | Sequence 1 | Sequence 2
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No